CLINICAL TRIAL: NCT04781101
Title: Can Robot-Assisted Gait Training In Addition To Conventional Rehabilitation Provide Better Outcomes In Terms Of Balance, Spasticity And Functionality In Children With Cerebral Palsy?
Brief Title: Can Robot-Assisted Gait Training In Addition To Conventional Rehabilitation Provide Better Outcomes In Children With Cerebral Palsy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13.02.2019-103
Record Dates: First submitted 2020-11-11; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy; Robotics
Keywords: Cerebral palsy; Robotics; Functional status
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional therapy (Experimental): conventional therapy
  Interventions: Other: conventional therapy
- RoboGait® (Experimental): Group 1 (n = 13) received conventional therapy (65 min, 2 days/week ×8) and group 2 (n = 13) received 25 minutes of robot-assisted gait training (RoboGait®) in addition to conventional therapy (40 min, 2 days/week ×8).
  Interventions: Other: RoboGait®

INTERVENTIONS:
Other: conventional therapy — Conventional therapy sessions that were planned by a physiotherapist for the children were conducted by a physiotherapist experienced in paediatrics. The therapy sessions mainly focused on functions such as the regulation of muscle tone, correction of posture, elimination of stiffness, muscle strengthening, balance/coordination training and mobilisation (Figure 2). The sessions were planned to last 40 minutes.
  Arms: conventional therapy
Other: RoboGait® — The RoboGait®-assisted gait system was used for the robot-assisted gait training. In addition to conventional therapy, 16 robot-assisted gait training sessions were conducted, each lasting 25 minutes for 2 days a week (400 minutes in total). Gait speed was 1.5 km/h in all sessions. Considering conditions such as joint limitations and spasticity, gait training was performed with patients bearing 45% to 75% of their weight.
  Arms: RoboGait®

SUMMARY:
A total of 26 patients who were diagnosed with CP [diplegic, with Gross Motor Function Classification System (GMFCS) level of 2-5] and who regularly participated in a rehabilitation programme were included in the study after obtaining approval from their parents. The patients were randomly assigned to two groups. Group 1 (n = 13) received conventional therapy (65 min, 2 days/week ×8) and group 2 (n = 13) received 25 minutes of robot-assisted gait training (RoboGait®) in addition to conventional therapy (40 min, 2 days/week ×8).

DETAILED DESCRIPTION:
Purpose: This study aimed to investigate the effects of robot-assisted training (RAT) on motor functions, spasticity status, balance and functionality in children with cerebral palsy (CP).

Method: A total of 26 patients who were diagnosed with CP [diplegic, with Gross Motor Function Classification System (GMFCS) level of 2-5] and who regularly participated in a rehabilitation programme were included in the study after obtaining approval from their parents. The patients were randomly assigned to two groups. Group 1 (n = 13) received conventional therapy (65 min, 2 days/week ×8) and group 2 (n = 13) received 25 minutes of robot-assisted gait training (RoboGait®) in addition to conventional therapy (40 min, 2 days/week ×8).

Outcome measures: GMFCS was used to evaluate motor functions and Modified Ashworth Scale was used to evaluate spasticity. Paediatric Berg Balance Scale, Paediatric Functional Independence Measure and timed up and go test were used to assess balance and functional status. The evaluations were performed at baseline and after 8 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

* diplegic CP and who were level 2-5 according to the Gross Motor Function Classification System (GMFCS) were included in the study. Children who presented with any disorder involving the peripheral nervous system or another neurological disorder such as epilepsy were not included.

Exclusion Criteria:

* Patients in whom the dose of their prescribed medication for spasticity was changed during the study period were excluded

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
GMFCS | 5 minute
  GMFCS was used to determine the extent and severity of CP in order to identify the inclusion criteria. The 5-level classification system that was developed in 1997 and expanded in 2007 by Palisano et al. was used to classify gross motor functions in patients with CP (7). The expanded Turkish version of GMFCS was prepared by Günel et al. (8). Levels of this classification are outlined below:
  Level I: Walks without limitations Level II: Walks with limitations Level III: Walks with the use of hand-held mobility equipment Level IV: Self-mobility is limited but can use a powered mobility device Level V: Carried on a manual 'wheelchair' GMFCS levels of children with CP were studied under 5 levels in this study. Children with CP who were level 2 and above were included
TUG test | 10 minute
  This test measures various components such as gait speed, postural control, functional mobility and balance (12). In the evaluation, a chair with a backrest but no armrests was placed at a 3-m distance from the wall and the children were positioned with hips and knees in 90° flexion. The children were asked to stand up, walk and touch the picture on the wall and then go back and sit down. The activity was shown and explained to the children before starting the test. Then, the children were asked to complete this activity twice. The time taken by the children to stand up from the chair, perform the activity and sit down was noted. The mean of the two test results was used for the analysis. Two children who were level 5 according to GMFCS were not included in this assessment.
WeeFIM | 20 minute
  WeeFIM was used to evaluate the level of functional skills in children with CP. It consists of 18 items in six domains including sphincter control, self-care, transfer, communication, locomotion, cognition and social interaction. Each item in these domains is scored from 1 to 7, considering whether the child is able to perform the relevant functional task in time with or without requiring a device or assistance. The item is scored 1 point if a child requires total assistance while performing the task and 7 if a child independently performs the task safely and in time. The items are scored from 1 to 7 depending on the requirement for assistance. Therefore, the lowest score is 18 (completely dependent) and the highest score is 126 (completely independent) (11).
PBBS | 15 minute
  PBBS, a modification of the Berg Balance Scale (BBS), developed for children by Franjoine et al. (10) was used to evaluate the functional balance of children during daily life activities. The scale consists of 14 items that are scored from 0 to 4, with a maximum score of 56 points. In PBBS, the order of the sections in the standard BBS has been rearranged from easy to difficult as a functional sorting, the time standards in the sections related to maintenance of static posture have been reduced considering the paediatric population and the guidance has been simplified (10).
Modified Ashworth Scale (MAS). | 15 minute
  MAS was used to evaluate the muscle tone of the gastrosoleus, gluteus medius and quadriceps femoris muscles in lower limbs. The children were allowed to rest on the therapy bed for 5 minutes before starting the assessment. The measurements were conducted on bare limbs at the same time of the day on a bed with suitable firmness and width, while the children were lying in the supine position with the upper and lower limbs placed parallel to the torso and in extension as much as possible and the head in middle position without a pillow. Passive range of motion exercises were conducted within 1 second for measurement standardisation purposes in MAS. The children included in the study were evaluated by the same physiotherapist.

CONTACTS AND LOCATIONS:
Overall Officials: Tülay Çevik Saldıran, PhD, Study Chair — Bitlis Eren University
Locations (1):
- Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No